CLINICAL TRIAL: NCT06561776
Title: Cough Strength, Physical Activity and Balance in Young Adults.
Brief Title: Investigation of Physical Impairments in Young Adults
Status: Recruiting | Type: Observational
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Gulsah Bargi, Principal Investigator, Izmir Democracy University
Other Study IDs: Young adults
Record Dates: First submitted 2024-08-16; First posted 2024-08-20 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Adult Children
Keywords: adult; balance; cough; COVID-19; physical activity
MeSH Terms: conditions — Cough; COVID-19; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Young adults: This group will consist of individuals aged 18 and over
  Interventions: Other: Physical Evaluations of individuals

INTERVENTIONS:
Other: Physical Evaluations of individuals — Participants will be evaluated on cough strength, physical activity and balance. The data to be obtained from all these evaluations are planned to be collected face to face from the participants at once and within a maximum of 1 hour.

SUMMARY:
Physical inactivity is widespread among young adults due to different disasters like the COVID-19 and earthquakes. On the other hand, it is unknown how physical activity level affects cough strength and balance in young adults. In current study, it was aimed to investigate both cough strength, physical activity and balance status in young adults and the relationship between these parameters.

DETAILED DESCRIPTION:
Participation in free time physical activities has various health benefits such as increasing academic success, improving quality of life. Physical inactivity in university students has been triggered by disasters such as COVID-19 and earthquakes that we have experienced. However, it is not yet known how physical inactivity and sedentary life affect cough strength and balance in these healthy young people. Thus, this study aimed to explore the cough strength, physical activity and balance status and the correlations between these parameters in young adults.

ELIGIBILITY:
Inclusion Criteria:

* being 18 years or older,
* volunteering to participate in the study
* understanding and answering the questionnaire

Exclusion Criteria:

* having any physical or mental disability/disease and/or cognitive impairment that would prevent physical activities
* being pregnant.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: At least 51 individuals aged 18 and over will be included
Sampling Method: Non-Probability Sample
Enrollment: 51 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Cough strength | through study completion, an average of 1 year
  Cough strength will be evaluated using a PEFmeter.

SECONDARY OUTCOMES:
Physical activity score | through study completion, an average of 1 year
  Physical activity will be assessed using the Short Form of International Physical Activity Questionnaire. There are a total of 7 questions in the questionnaire. It provides a total physical activity score. As this score increases, physical activity level of the participant increases.
Static balance score | through study completion, an average of 1 year
  It was assessed with a single-leg balance test and the maximum time in this position was recorded in seconds with a stopwatch.
Dynamic balance score | through study completion, an average of 1 year
  I was assessed with the standing functional reach test. Participant was asked to extend their arms forward parallel to the wall, the distance between the starting point and the farthest reached point was measured. As this distance increases, the balance increases.

CONTACTS AND LOCATIONS:
Overall Officials: GÜLŞAH BARĞI, Study Director — Izmir Democracy University; ALPEREN BİNİCİ, Principal Investigator — Izmir Democracy University; GÖKAY GÖKÇE, Principal Investigator — Izmir Democracy University; MAHİR SOLMAZ, Principal Investigator — Izmir Democracy University; BİLAL KAMACİHAN, Principal Investigator — Izmir Democracy University
Locations (1):
- Izmir Democracy University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Silva MVGD, Soares IC, Ventura SC, Kuroda MN, Goncalves Dos Santos BG, Nogueira da Silva C, Borato LA, Pedroni CR. Trunk muscles influence lower limb performance in crossfit athletes: A cross-sectional study. Physiother Res Int. 2024 Jan;29(1):e2040. doi: 10.1002/pri.2040. Epub 2023 Jul 15. PMID 37452583
- [Background] Koca R, Sen ME. The effect of anthropometric measurements and muscle endurance of the trunk and lower extremities on anatomic body awareness in healthy individuals with different levels of physical activity. Acta Neurol Belg. 2024 Jun;124(3):995-1003. doi: 10.1007/s13760-024-02526-9. Epub 2024 Mar 28. PMID 38546933